CLINICAL TRIAL: NCT00634114
Title: A Multicentre, Randomised, Double-blind, Parallel-group, Comparative Study to Compare the Efficacy and Safety of Esomeprazole 20 mg Once Daily Oral Administration With Omeprazole 10 mg and Esomeprazole 10 mg Once Daily Oral Administration in Maintenance Treatment in Patients With Healed Reflux Esophagitis
Brief Title: Reflux Esophagitis Phase III Study (Maintenance Treatment)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind / Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D961HC00006
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Results first posted 2010-06-17 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-05

CONDITIONS: Reflux Esophagitis
Keywords: Reflux Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Esomeprazole; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Esomeprazole and Omeprazole
  Interventions: Drug: Esomeprazole; Drug: Omeprazole
- 2 (Experimental): Esomeprazole
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — 10mg once daily oral administration
  Other Names: Nexium
  Arms: 1
Drug: Esomeprazole — 20mg once daily oral administration
  Other Names: Nexium
  Arms: 2
Drug: Omeprazole — 10mg once daily oral administration
  Other Names: Prilosec
  Arms: 1

SUMMARY:
The primary objective of this study is to evaluate the efficacy of esomeprazole 20 mg once daily for 24 weeks on maintenance of Reflux Esophagitis in patients with healed reflux esophagitis in comparison with omeprazole 10 mg once daily and esomeprazole 10 mg once daily by assessment of presence/absence of recurrence of Reflux Esophagitis throughout the treatment period (from the randomisation to the treatment completion) according to the Los Angeles classification.

ELIGIBILITY:
Inclusion Criteria:

* Patients with healed Reflux Esophagitis verified by EGD in the preceding study (D961HC00002)
* Patients with endoscopically verified healed Reflux Esophagitis by EGD receiving general treatment with PPI

Exclusion Criteria:

* Gastric or duodenal ulcer verified by EGD within 12 weeks before randomisation.
* Use of any PPI from 14 days before EGD performed at the screening visit to the day of randomisation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2008-01; Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maotsugu Oyama, MD, PhD, Study Director — AstraZeneca
Locations (44):
- Japan (44):
  - Research Site, Akita, Akita
  - Research Site, Kashiwa, Chiba
  - Research Site, Kisarazu, Chiba
  - Research Site, Kōriyama, Fukishima
  - Research Site, Nihonmatsu, Fukishima
  - Research Site, Nishishirakawa, Fukishima
  - Research Site, Fukuoika, Fukuoka
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kurume, Fukuoka
  - Research Site, Nukaya, Fukuoka
  - Research Site, Fukuoka, Fukuolka
  - Research Site, Kōriyama, Fukushima
  - Research Site, Shirakawa, Fukushima
  - Research Site, Sugawa, Fukushima
  - Research Site, Gifu, Gifu
  - Research Site, Maebashi, Gunma
  - Research Site, Yasunaka, Gunma
  - Research Site, Sapporo, Hokkaido
  - Research Site, Hitachi, Ibaraki
  - Research Site, Mito, Ibaraki
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Sakaidechō, Kagawa-ken
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Fujisawa, Kanagawa
  - Research Site, Kawasaki, Kanagawa
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Shibata, Myagi
  - Research Site, Kiso, Nagano
  - Research Site, Matsumoto, Nagano
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Fujiidera, Osaka
  - Research Site, Toyonaka, Osaka
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Ohtawara, Tochigi
  - Research Site, Toshima-ku, Tokayo
  - Research Site, Adachi City, Tokyo
  - Research Site, Hachiōji, Tokyo
  - Research Site, Kiyose, Tokyo
  - Research Site, Setagaya City, Tokyo
  - Research Site, Shinagawa, Tokyo
  - Research Site, Tottori-shi, Tottori
  - Research Site, Shimonoseki, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolment 8Jan08-19May09. 564 randomised participants, 563 in Full Analysis set and safety analysis set. FAS used for summaries of baseline characteristics and efficacy. SAS for summaries of safety. 1 pt. in Omep. 10 mg excluded as they took no investigational drug. Nos. for gender were 188 in Esom. 20 mg, 188 in Esom. 10 mg and 187 in Omep. 20 mg.
Pre-assignment Details: Out of 578 enrolled participants, 564 participants were randomised and 14 participants were not randomised. The reasons of no randomisation were 'Incorrect enrolment' (11 participants) and 'Voluntary discontinuation by participant' (3 participants).
Groups:
- Experimental: Esomeprazole 20 mg: Esomeprazole 20 mg once daily
- Experimental: Esomeprazole 10 mg: Esomeprazole 10 mg once daily
- Comparator: Omeprazole 10 mg: Omeprazole 10 mg once daily
Period: Overall Study
Arm/Group | Experimental: Esomeprazole 20 mg | Experimental: Esomeprazole 10 mg | Comparator: Omeprazole 10 mg
Started | 188 (Randomised) | 189 (Randomised) | 187 (Randomised)
Completed | 160 (Completed) | 154 (Completed) | 148 (Completed)
Not Completed | 28 | 35 | 39
Not completed — Adverse Event | 6 | 8 | 3
Not completed — Withdrawal by Subject | 9 | 6 | 11
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 3 | 3 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Incorrect enrolment | 0 | 1 | 0
Not completed — Recurrence of reflux esophagitis | 5 | 15 | 21
Not completed — Difficult to continue | 3 | 1 | 1
Not completed — Other reason | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Esomeprazole 20 mg | Experimental: Esomeprazole 10 mg | Comparator: Omeprazole 10 mg | Total
Number analyzed (Participants) | 188 | 189 | 187 | 564
Age, Customized [Number; unit: Participants]
  <65 | 131 [131 to NA] | 131 [131 to NA] | 137 [137 to NA] | 399 [0 to 0]
  65-74 | 45 [45 to NA] | 41 [41 to NA] | 38 [38 to NA] | 124 [0 to 0]
  >=75 | 12 [12 to NA] | 16 [16 to NA] | 12 [12 to NA] | 40 [0 to 0]
  Missing | 0 [0 to NA] | 1 [1 to NA] | 0 [0 to NA] | 1 [0 to 0]
Sex/Gender, Customized [Number; unit: Participants] — 1 participant was excluded in Esomeprazole 10 mg as they did not take any investigational drug.
  Participants
    Female | 46 [142 to NA] | 51 [137 to NA] | 42 [145 to NA] | 139 [0 to 0]
    Male | 142 [46 to NA] | 147 [51 to NA] | 145 [42 to NA] | 434 [0 to 0]
    Missing | 0 [0 to NA] | 1 [1 to NA] | 0 [0 to NA] | 1 [0 to 0]

OUTCOME MEASURES:

1. Secondary Outcome: Absence of Recurrence of Reflux Esophagitis According to Los Angeles Classification up to 4 Weeks After Treatment
Description: Los Angels classification consists of 5 grades (Grade O, Grade A, Grade B, Grade C and Grade D). A patient classfied into Grade O was considered no reflux esophagitis. The participants who had a healing of reflux esophagitis with Grade O at Visit 1 were randomised. Number of participants who did not have Grades A-D up to 4 weeks after treatment was evaluated.
Time Frame: up to 4 weeks
Measure: Number; unit: Participants
Arm/Group | Experimental: Esomeprazole 20 mg | Experimental: Esomeprazole 10 mg | Comparator: Omeprazole 10 mg
Number analyzed (Participants) | 188 | 188 | 187
Participants | 184 | 180 | 171

2. Primary Outcome: Absence of Recurrence of Reflux Esophagitis According to Los Angeles Classification Throughout the Treatment Period.
Description: Los Angels classification consists of 5 grades (Grade O, Grade A, Grade B, Grade C and Grade D). A patient classfied into Grade O was considered no reflux esophagitis. The participants who had a healing of reflux esophagitis with Grade O at Visit 1 were randomised. Number of participants who did not have Grades A-D throughout the treatment period was evaluated.
Time Frame: Up to 24 weeks
Measure: Number; unit: Participants
Arm/Group | Experimental: Esomeprazole 20 mg | Experimental: Esomeprazole 10 mg | Comparator: Omeprazole 10 mg
Number analyzed (Participants) | 188 | 188 | 187
Participants | 174 | 166 | 156

3. Secondary Outcome: Absence of Recurrence of Reflux Esophagitis According to Los Angeles Classification up to 12 Weeks After Treatment
Description: Los Angels classification consists of 5 grades (Grade O, Grade A, Grade B, Grade C and Grade D). A patient classfied into Grade O was considered no reflux esophagitis. The participants who had a healing of reflux esophagitis with Grade O at Visit 1 were randomised. Number of participants who did not have Grades A-D up to 12 weeks after treatment was evaluated.
Time Frame: Up to 12 weeks
Measure: Number; unit: Participants
Arm/Group | Experimental: Esomeprazole 20 mg | Experimental: Esomeprazole 10 mg | Comparator: Omeprazole 10 mg
Number analyzed (Participants) | 188 | 188 | 187
Participants | 179 [NA to NA] | 172 [NA to NA] | 163 [NA to NA]

ADVERSE EVENTS:
Description: 1 participant was excluded in Esomeprazole 10 mg as they did not take any investigational drug.
Arm/Group | Experimental: Esomeprazole 20 mg | Experimental: Esomeprazole 10 mg | Comparator: Omeprazole 10 mg
Serious Adverse Events (participants affected / at risk) | 5/188 | 4/188 | 1/187
Other Adverse Events (participants affected / at risk) | 71/188 | 69/188 | 34/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Esomeprazole 20 mg (N=188) | Experimental: Esomeprazole 10 mg (N=188) | Comparator: Omeprazole 10 mg (N=187)
Colonic polyp (Gastrointestinal disorders) | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Esomeprazole 20 mg (N=188) | Experimental: Esomeprazole 10 mg (N=188) | Comparator: Omeprazole 10 mg (N=187)
Nasopharyngitis (Infections and infestations) | 31 | 37 | 31
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 11 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 7 | 7
Gastric polyps (Gastrointestinal disorders) | 3 | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 5
Constipation (Gastrointestinal disorders) | 2 | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 4
Blood creatine phosphokinase increased (Investigations) | 5 | 5 | 2
Blood pressure increased (Investigations) | 1 | 5 | 1
Contusion (Injury, poisoning and procedural complications) | 5 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study withiout AZ approval before this study was completed.